CLINICAL TRIAL: NCT01702818
Title: Stress Hormones, Mood and Women's Sexual Desire (MODEST)
Acronym: MODEST
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Lori Brotto, Associate Professor, University of British Columbia
Other Study IDs: H10-02067
Record Dates: First submitted 2012-08-27; First posted 2012-10-08 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2017-05

CONDITIONS: Hypoactive Sexual Desire Disorder (HSDD)
Keywords: Hypoactive Sexual Desire Disorder; HSDD; Cortisol; DHEA; Stress Hormones; Sexual Desire; Mood; Sexual Function; Childhood Maltreatment; Childhood Abuse
MeSH Terms: conditions — Sexual Dysfunctions, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — saliva samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HSDD group: Women with a diagnosis of Hypoactive Sexual Desire Disorder (HSDD).
- Control Group: Women without a diagnosis of Hypoactive Sexual Desire Disorder (HSDD).

SUMMARY:
Women with Hypoactive sexual desire disorder (HSDD) have all measures of testosterone activity comparable to controls but lower levels of dehydroepiandrosterone (DHEA). Although DHEA is a precursor of testosterone it has other actions including involvement in the stress system. It is also linked to mood. This study focuses on measures of childhood stress, current mood and salivary stress hormones, in women with and without HSDD. We hypothesize that low levels of DHEA reflect dysfunction of the neuroendocrine stress response system involving the brain, pituitary and adrenal glands where DHEA is produced.

ELIGIBILITY:
Inclusion Criteria for HSDD Group:

* (1) diagnosis of HSDD
* (2) over 19 years of age
* (3) sexual complaints of low desire of at least 12 months duration.

Inclusion criteria for Control group:

* (1) sexually healthy, i.e., must not meet criteria for any sexual dysfunction, as determined by a telephone screening, followed by an in-person structured assessment, the Decreased Sexual Desire Screener (DSDS)
* (2) over 19 years of age.

Exclusion Criteria for both Control and HSDD groups:

* (1) lack of fluency in English
* (2) currently meeting DSM-IV-TR diagnostic criteria for major depressive disorder as measured by an in-person, semi-structured interview based on the Major Depressive Disorder Module of the Structured Clinical Interview for DSM-IV-TR (SCID-I
* (3) current use of prescription drugs such as antidepressants or other medications with known sexual side effects (e.g., glucocorticoids, aromatase inhibitors), or known effects on cortisol metabolism, or use of illicit drugs
* (4) use of hormone replacement therapy or hormonal contraceptives;
* (5) a body mass index (BMI) <18.5 or >29.9
* (6) cigarette smoking
* (7) chronic medical or psychiatric disease with potential to interfere with sexual function (e.g., chronic neurological disease, cardiac and liver disease, eating disorders, anxiety disorders)
* (8) chronic pain with intercourse not relieved by a vaginal lubricant
* (9) loss of genital responsiveness
* (10) significant relationship discord
* (11) not having a family physician who we could contact if depression is diagnosed during the assessment
* (12) difficulty in complying with questionnaires or in completing interview.

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with and without a diagnosis of Hypoactive Sexual Desire Disorder (HSDD).
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2012-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
DHEA levels | Data is collected at 4 time points on 3 separate days
  DHEA levels derived from saliva samples.

SECONDARY OUTCOMES:
Cortisol levels | Data is collected at 4 time points on 3 separate days
  Cortisol levels derived from saliva samples.
Depression | data is collected at single time point
  Depression will be measured by the Beck Depression Inventory (Beck & Beamesderfer, 1974)
Perceived stress | data is collected at a single time point
  Perceived stress will be measured with the 10-item Perceived Stress Scale (Roberti, Harrington & Storch 2006)
Sexual function | data is collected at a single time point
  Self-report sexual function will be measured with the Sexual Interest and Desire Inventory (Clayton et al. 2006))
Relationship satisfaction | data is collected at a single time point
  Relationship satisfaction will be measured with the Relationship Assessment Scale (Hendrick, 1988) and the Dyadic Adjustment Scale (Spanier, 1976)
History of childhood trauma | dat is collected at a single timepoint
  History of childhood trauma will be determined with the Childhood Trauma Questionnaire (Bernstein & Fink, 1995)
History of childhood sexual abuse | data is collected at a single time point
  History of Childhood Sexual Abuse will be determined with the Childhood Sexual Abuse Measure (Finkelhor, 1979)
PTSD symptoms | data is collected at a single time point
  Presence and severity of post traumatic stress disorder symptoms will be determined through the Clinician-Administered PTSD Scale (Blake et al. 1998)

CONTACTS AND LOCATIONS:
Overall Officials: Rosemary Basson, MD, Principal Investigator — University of British Columbia; Lori A Brotto, PhD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Centre for Sexual Medicine, Vancouver, British Columbia, Canada

REFERENCES:
- See also: UBC Sexual Health Lab — http://brottolab.med.ubc.ca/